CLINICAL TRIAL: NCT00262210
Title: A Comparative Study for Non-Hodgkin's Lymphoma in Hepatitis B Virus Carriers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1495
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2005-12-06 (Estimated); Status verified 2005-12

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: Cyclophosphamide Epirubicin Etoposide Prednisolone

SUMMARY:
* AIMS OF THE STUDY

1. To test if steroid-free chemotherapeutic regimens decrease the risk of HBV reactivation and hepatitis development in HBsAg (+) carriers.
2. To compare the efficacy of steroid-free chemotherapeutic regimens with that of steroid-containing regimens in terms of lymphoma control.
3. To study the change of activity of HBV and other hepatotropic viruses during the course of chemotherapy.

DETAILED DESCRIPTION:
* TREATMENT PLANS FOR FIRST-LINE AND SECOND LINE CHEMOTHERAPY

1. First-line Chemotherapy 1.1 PACE and ACE Treatment Scheme of PACE and ACE* Cyclophosphamide 650 mg/m2, i.v. Day 1 Epirubicin 60 mg/m2, i.v. Day 1 Etoposide 55 mg/m2/d, i.v. Day 1-3 Prednisolone 60 mg/m2/d, p.o. Day 1-7

   * For ACE, prednisolone is omitted. 1.2 Courses will be repeated every 21 days. 1.3 For patients with CR, give at least 2 additional courses for a minimum of 6 courses.

   1.4 For patients with PR or SD, may change to second-line chemotherapy if no further tumor shrinkage between two consecutive courses.Local radiotherapy is allowed for residual localized tumors.

   1.5 For patients with PD, change to second-line chemotherapy .
2. Second-line Chemotherapy : For patients who have failed steroid-containing or steroid- free chemotherapy, respective steroid-containing and steroid-free salvage chemotherapy should be used.

2.1 VIMP and VIM Treatment Scheme of VIMP and VIM* VP-16 100 mg/m2/d, i.v. Day 1,3,5 Ifosfamide 1 gm/m2/d, i.v. Day 1-5 MTX 30 mg/m2/d, i.v. Day 1,5 Prednisolone 60 mg/m2/d, P.O. Day 1-7

* For VIM, prednisolone is omitted. Repeated every 21 days.

Mesna for urinary tract protection is needed:

Mesna 100 mg/m2 is bolus injected immediately before the infusion of first-day ifosfamide, and then 500mg/m2/day is infused for 5 day with ifosfamide.

2.2 Infusional CDE + P (ICDE + P) and Infusional CDE (ICDE) Treatment Scheme of ICDE+P and ICDE* Cyclophosphamide 187.5 mg/m2/d, continuous i.v. infusion Day 1-4 Epirubicin 20 mg/m2/d, continuous i.v. infusion Day 1-4 Etoposide 60 mg/m2/d, continuous i.v. infusion Day 1,4 Prednisolone 60 mg/m2/d, P.O. Day 1-7

* For ICDE, prednisolone is omitted. Repeated every 21 days.

  * Cyclophosphamide and epirubicin can be mixed in a 500ml of 5% D/W, and infused together. Etoposide is dissolved in another 500ml of 5% D/W, and infused in a separate line.

3.0 DOSE MODIFICATION 3.1 Hematological Toxicity*

Drug administration is postponed one week if there is no full hematological recovery (AGC > 2,000/mm3 and Platelet > 100,000/mm3 ) from prior course at scheduled treatment day. Full doses will be given as soon as the hematological recovery is documented. If after another one week, i.e. two weeks after the due day, recovery is still incomplete, the treatment may be started and the dosage of the drugs be reduced according to the following schedule for all regimens:

AGC*/mm3Platelet/mm3 1,500-2,00075,000-100,000 1,000-1,49950,000-74,999 <1,000<50,000 Cyclophosphamide 80% 60% ** Epirubicin 80% 60% ** VP-16 80% 60% ** Ifosfamide 80% 60% ** MTX 80% 60% **

* Growth factors (G-CSF, GM-CSF) are allowed to be used for patients with prolonged myelosuppression, but should not influence the schedule of dose- modification as illustrated above.

  * Postpone for another week. If the counts remain AGC < 1000 or Platelet < 50,000, growth factors may be used at this juncture, i.e. 2 weeks after due day. Patients should be off study if still AGC < 1,000 or Platelet < 50,000, 3 weeks after the due day.

3.2 Hepatotoxicity For patients with normal or abnormal prechemotherapy serum ALT, hepatitis or hepatitis flare-up is defined as a threefold or greater increase in serum ALT level that exceeds 100 IU/L. The hepatitis or hepatitis flare-up is attributed to reactivation of chronic hepatitis B when there is a sudden elevation (> 10-fold) in serum HBV DNA level or reappearance of HBV DNA or HBeAg in the serum.

Since serum HBV DNA data is not readily available in most hospitals, all patients with hepatitis or hepatitis flare-up are considered as HBV reactivation until proved otherwise. Cross-over to steroid-free arm for subsequent treatment is not allowed in this study. For patients with only minor hepatic dysfunction (Total Bilirubin <3.0 mg/dl and ALT <200 I.U./L), full-dose chemotherapy is recommended on the scheduled treatment date without delay. For patients with more severe hepatic dysfunction (total bilirubin ≧ 3.0 mg/dl or ALT ≧ 200 I.U./L), subsequent course is postponed for 1 week and the dosage modified as followings if the values remain abnormal after 1 week:

Total Bilirubin (mg/dl) <3.0 3.0 - 4.9 5.0 - 7.5 >7.5 ALT (I.U./L) <200 200 - 399 400 - 800 >800 Epirubicin 100% 75% 50% *

* Wait until recovery with serum levels below these values. Patients will be off study if Bil > 7.5 or ALT > 800, 3 weeks after the due day.

3.3 Gastrointestinal Toxicity In case of severe (≧ ECOG grade III) anorexia, nausea, vomiting, diarrhea, stomatitis or abdominal pain, all therapy should be delayed until improvement of symptoms to ≦ GrII.

Patient will be off study if ≧ GrIII toxicity persists ≧ 3 weeks after due day. Patients are allowed to use H3-blockers in the subsequent courses for severe nausea and vomiting. If gastrointestinal toxicity is still ≧ Gr II during the next course, doses of cyclophosphamide, epirubicin and VP-16 should be reduced by 25% in the subsequent courses. If no further episodes of severe reaction, the doses can be escalated back to 100%.

3.4 Cardiotoxicity In case of ECOG grade II cardiotoxicity, epirubicin should be reduced by 50%. If cardiotoxicity resolved, the dose may be carefully escalated i.e., increase 10-25% of dose each time, in the subsequent courses. If severe (≧ ECOG grade III) cardiotoxicity develops, epirubicin should be discontinued and should not be used again in the subsequent courses.

3.5 In the event of multiple toxicities, dose modification should be made based on the guideline that requires the greatest reduction of doses.

4. CRITERIA FOR REMOVAL FROM STUDY

All patients who are still under or have completed protocol treatments (1st-line or 2nd-line) should be continuously followed-up for all study end points. Patients are removed from study if they have major violation of the protocol due to the following reasons:

4.1 Refuse treatment. 4.2 Unable to receive due treatments either because of severe toxicity or other reasons.

4.3 Inadvertent cross-over to opposite arms (steroid-containing or steroid-free) of treatment.

ELIGIBILITY:
* Inclusion Criteria:

  1. Histologically proven NHL, and for which intensive chemotherapy is considered treatment-of-choice.
  2. HBsAg-positive.
  3. No previous chemotherapy and radiotherapy.
  4. No concurrent radiotherapy. AGC ≧ 2,000/mm3, Platelet ≧ 100,000/mm3 of peripheral blood.
  5. Total bilirubin ≦ 2.5 mg/dl. Alanine aminotransferase (SGPT) < 200 I.U/L
  6. Serum creatinine ≦1.5 mg/dl Blood urea nitrogen (BUN) ≦ 25 mg/dl
  7. Objectively measurable or evaluable disease
  8. Signed informed consent
* Exclusion Criteria:

  1. Age > 75 years, or Age < 15 years
  2. Pregnant or breast-feeding women.
  3. Patients with history of brain metastasis or CNS involvement.
  4. Child's class B or C in patients with liver cirrhosis.
  5. Impaired cardiac function with NYHA (New York Heart Association) classification ≧ GrII.
  6. Concurrent glucocorticoids use (for other reasons). The conventional use of glucocorticoids for antiemetic purpose is also not allowed.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1995-06; Study Completion 1999-12

PRIMARY OUTCOMES:
We expect to enter 25 patients per year and finish accrual of patients within 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, Ph.D., Principal Investigator — Lymphoma Disease Committee of TCOG
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan